CLINICAL TRIAL: NCT06620146
Title: The Short-Term and Long-Term Effects of Providing Mechanical Bath in Terminally Ill Patients: A Randomized Controlled Trial
Brief Title: The Short-Term and Long-Term Effects of Providing Mechanical Bath in Terminally Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202207077RINB
Record Dates: First submitted 2024-09-22; First posted 2024-10-01 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2022-08

CONDITIONS: Hospice and Palliative Care Nursing; Terminally Ill Patients
Keywords: mechanical bathing; instrument validation; hospice care; comfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group provided with mechanical bathing every other day for a week (Experimental): Participants in the intervention group will be provided mechanical bathing every other day for a week.
  Interventions: Other: mechanical bathing
- control group provided with routine care (mechanical bathing once a week) (No Intervention): control group receive routine care (using mechanical bathing once a week)

INTERVENTIONS:
Other: mechanical bathing — Providing mechanical bathing (MB) is a commonly used strategy to maintain cleanness and comfort in patients with terminally illness. The electric medical bathtub (ARJO, Rhapsody) provides functions such as showering, bathing, and water massage. The MB will be operated by 2-3 nursing staff, trained hospice volunteers, or researchers. Each patient's MB process lasts about 20 minutes, including washing the hair and body with a handheld showerhead, followed by soaking in warm water for about 5-10 minutes. Based on the patient preference, the water temperature is adjusted between 38 to 40 degrees Celsius.
  Arms: intervention group provided with mechanical bathing every other day for a week

SUMMARY:
Providing mechanical bathing (MB) is a commonly used strategy to maintain cleanness and comfort in patients with terminally illness. However, extra devices, costs, and human resources are required for such service. There is also a lack of evidence systematically examining the benefits of using MB. These extra financial and resource burden and insufficient evidence limit the use of MB in hospice clinical settings. The aim of this study is to examine whether more frequent MB can improve hospice patients' and their caregivers' comfort. The study has two phases. The first preparation phase is for questionnaire translation and piloting. The second phase is a randomized controlled trail in which adult hospice patients admitted to a hospice unit will be randomly assigned to intervention or control group. Participants in the intervention group will be provided MB every other day for a week while participants in the control group receive routine care (using MB once a week). The primary outcome is patients' level of comfort as measured by questionnaire and physical indicators. The secondary outcome is caregivers' emotional burden. Data collection will occur before, during, and after the intervention. The estimation sample sizes for the two phases are 200-250 and 80, respectively. Descriptive analysis and generalized estimating equations will be employed to analyze data. The results of this study will fully recognize the short-term and long-term effects of MB. This understanding can then serve as a foundation to standardize the frequency of providing MB and justify for the resources needed for providing MB.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Diagnosed by a physician as having a terminal illness and currently receiving treatment in the palliative care unit of National Taiwan University Hospital
* Unable to clean oneself
* Willing to receive MB
* Has not received any MB during this hospital stay
* If the caregiver will be responsible for caring for the patient throughout the study period, will also be invited to participate in the study

Exclusion Criteria:

* The patient, due to physical, consciousness, or cognitive impairments, is unable to self-assess their symptoms, and there is no primary caregiver available during the study period to assist in evaluating their symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Physical comfort part-1 | Data collection occurs at four points: baseline (within 1 week after admission, before first MB), T1 (within 2 hrs after second MB), T2 (within 2 hrs after third MB), and T3 (one week after baseline).
  Physical comfort part-1 scale is assessed by two domains, including vital signs and pitting edema level. Vital signs contains temperature, heart rate, respiratory rate and blood pressure. Pitting edema is evaluated by grade +1 to +4, higher score means significant level of edema.
Physical comfort part-2 | Data collection occurs at two points: baseline (within 1 week after admission, before first MB) and T3 (one week after baseline).
  Physical comfort part-2 is assessed by pain and infection incidence. In the pain assessment, numerical rating scale and analgesic usage are for subjective and objective pain, respectively. Infection incidence is identified by new positive cultures, fever with a suspected source, new antibiotics, or abnormal markers such as C-reaction protein, white blood cell count and procalcitonin.
Agitation | Data collection occurs at four points: baseline (within 1 week after admission, before first MB), T1 (within 2 hrs after second MB), T2 (within 2 hrs after third MB), and T3 (one week after baseline).
  Agitation is assessed by Richmond Agitation Sedation Scale, which abbreviated as RASS, grading from -5 to +4, zero point means alert but calm. Higher scores means intense agitation and lower scores means stupor/drowsiness.
Physiological and psychological comfort | Data collection occurs at four points: baseline (within 1 week after admission, before first MB), T1 (within 2 hours after second MB), T2 (within 2 hours after third MB), and T3 (one week after baseline).
  Physiological and psychological comfort is assessed by symptoms (Edmonton Symptom Assessment System, ESAS), which have 11 items including physical and mental that grading from 1 to 10 points of each question. Higher scores means more symptoms.
Psychospiritual, sociocultural and environmental comfort | Data collection occurs at four points: baseline (within 1 week after admission, before first MB), T1 (within 2 hrs after second MB), T2 (within 2 hrs after third MB), and T3 (one week after baseline).
  Psychospiritual comfort is measured by the Hospice Comfort Questionnaire (HCQ), which have 24 items rating from 1 to 6 points of each question, higher level means less uncomfortable. Moreover, the HCQ assessment also covers sociocultural and environmental comfort.

SECONDARY OUTCOMES:
Emotional burden of family members | Data was collected at two points: baseline (within 1 week after admission, before first MB) and T3 (one week after baseline).
  Emotional burden of family members, will be measured using the Mood Thermometer (Brief Symptom Rating Scale, BSRS-5), rating from 0-4 points of each item. A higher total score of BSRS-5 indicates a higher emotional burden of the family member.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No